CLINICAL TRIAL: NCT04969497
Title: A Randomized Open-Label Three-Way Crossover Study to Compare the Pharmacokinetics, Safety, and Tolerability of Two Lots of M207 3.8 mg (Administered as Two 1.9 mg Patches on the Upper Arm for 30 Minutes) and Intranasal Zolmitriptan 5.0 mg x 2 Doses in Healthy Volunteers
Brief Title: Study of PK, Safety, and Tolerability of 2 Lots of M207 & Intranasal Zolmitriptan in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-2021-001
Record Dates: First submitted 2021-06-28; First posted 2021-07-20 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Migraine
Keywords: Pharmacokinetics; Healthy; Volunteer
MeSH Terms: conditions — Migraine Disorders | interventions — zolmitriptan

STUDY DESIGN:
Intervention Model Description: Subjects are randomized to receive one of six treatment sequences of three open-label treatments 48 hours apart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence ABC (Experimental): Receives interventions in the sequence, A, B, C.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
- Sequence CAB (Experimental): Receives interventions in the sequence, C, A, B.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
- Sequence BCA (Experimental): Receives interventions in the sequence, B, C, A.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
- Sequence CBA (Experimental): Receives interventions in the sequence, C, B, A.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
- Sequence BAC (Experimental): Receives interventions in the sequence, B, A, C.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
- Sequence ACB (Experimental): Receives interventions in the sequence, A, C, B.
  Interventions: Drug: Treatment A: M207 3.8 mg "MiniMac"; Drug: Treatment B: M207 3.8 mg "MACAP"; Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0

INTERVENTIONS:
Drug: Treatment A: M207 3.8 mg "MiniMac" — Treatment A: M207 3.8 mg administered as two 1.9 mg patches 30 minutes wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups
  Other Names: MiniMac; M207
Drug: Treatment B: M207 3.8 mg "MACAP" — Treatment B: M207 3.8 mg administered as two 1.9 mg patches 30 minutes wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups
  Other Names: MACAP; M207
Drug: Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0 — Treatment C: 5.0 mg Intranasal Zolmitriptan administered at time = 0 and 2 hours post time 0
  Other Names: Zomig

SUMMARY:
This is a single-center, open-label, randomized, 3-way crossover study. Each subject will receive each of the three study treatments once, followed by in-clinic monitoring and extensive blood sample collection for plasma PK analysis.

Dosing will occur at least 48 hours apart from the time of patch application, until completion of dosing in randomized order per the treatment sequence schedule. After completion dosing, subjects will be assessed one final time.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, three-way crossover study. Each subject will receive each of the three study treatments once, followed by in-clinic monitoring and extensive blood sample collection for pharmacokinetic analysis.

Dosing will occur at least 48 hours apart from the time of patch application, until completion of dosing in randomized order per the treatment sequence schedule. Subjects may be dosed in 2 or more separate groups in each period, for example, 24 subjects on one day and 24 subjects on another day.

Plasma samples from the dosing days will be sent to the analytical laboratory for analysis. Tolerability scores for each of the dose levels will be summarized.

After completion of the three dosing days, subjects will be assessed one final time and dismissed from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men 18 to 50 years of age (inclusive)
2. Good general health with no clinically significant abnormalities as determined by medical history, physical examination, CBC, blood chemistry, urinalysis, and ECG.
3. Negative serum pregnancy tests (for female subjects) at the screening and admission visit.
4. Consent of female subjects to use a medically effective method of contraception throughout the entire study period and for 30 days after the subject completes the study. Medically effective methods of contraception that may be used by the subject include abstinence, use of diaphragm and spermicide, intrauterine device (IUD), rings, condom and vaginal spermicide, non-oral hormonal contraceptives (subjects must be stable on non-oral hormonal contraceptives for at least 3 months prior to screening), surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy, hysteroscopic sterilization) and post-menopausal (≥ 2 years of amenorrhea).
5. Ability to read, understand, and provide written informed consent that they understand the purpose of the study and procedures required for the study before enrolling in the study, and willingness to comply with all study procedures and restrictions.

Exclusion Criteria:

1. Evidence of significant history of hepatic, reproductive, gastrointestinal, renal, bleeding, or hematological disorders including coagulation, pulmonary, neurological, respiratory, endocrine, or cardiovascular system abnormalities (especially hypertension, peripheral vascular disease, coronary artery disease, transient ischemic attacks, or cardiac rhythm abnormalities), psychiatric disorders, acute infection, or other conditions that would interfere with study participation or with the absorption, distribution, metabolism, or excretion of drugs.
2. Presence of three or more of the following CAD risk factors for cardiovascular disease:

   A. Current tobacco use (subjects who have smoked within 30 days of screening) B. Hypertension (systolic BP > 140 or diastolic BP > 90) or receiving anti-hypertensive medication for treatment of hypertension C. Hyperlipidemia - LDL > 159 mg/dL and/or HDL < 40 mg/dL (or on prescribed anti-cholesterol treatment) D. Family history of premature coronary artery disease (CAD) (< 55 years of age in male first-degree relatives or < 65 years of age in female first degree relatives) E. Diabetes mellitus
3. Any contraindication to zolmitriptan administration including:

   * History of coronary artery disease or coronary vasospasm
   * Symptomatic Wolf-Parkinson-White syndrome or other cardiac accessory conduction pathway disorders
   * History of stroke, transient ischemic attack, or hemiplegic or basilar migraine
   * History or current Peripheral Vascular Disease
   * History or current Ischemic bowel disease
   * Hypertension (greater than or equal to 140/90 mmHg at either the screening or admission/baseline visit
   * Any history of hepatic impairment defined as ALT > 150 U/L, AST > 130 U/L or bilirubin > 2 times the ULN
4. History of contact dermatitis or known dermatological disorders that would interfere with the study procedures or assessments
5. Planned participation in activities which cause inflammation, irritation, sunburn, lesions, or tattoos at the intended application sites from 2 weeks prior to dosing through the duration of the trial
6. Use of any prescription anticoagulant within 30 days prior to the first dose through the duration of the trial
7. Use of prescription and over the counter medications within one week of dosing other than the following:

   * Hormone Replacement Therapy (HRT)
   * Non-oral hormonal birth control such as patches, IUD, rings, injections, or implants (all non-oral hormonal contraceptives) are allowed provided the dose has been stable for at least three months prior to screening and may be continued throughout the study
   * Antihistamines
   * Intermittently used NSAIDS
   * Acetaminophen if medically necessary (not more than 1000 mg/day)
8. Current known allergy or sensitivity to zolmitriptan or its derivatives or formulations
9. Current known allergy or sensitivity to tapes or adhesives
10. Use of any other investigational compound within 30 days of planned study drug dosing
11. Current use or history of drug and/or alcohol abuse within 6 months of screening and deemed to be clinically significant by the investigator
12. History of nasal pathology (e.g., polyps, significant septal deviation or perforation) or abnormal nasal exam (with findings such as nose piercing, gross deformities, and/or severe congestion) deemed to be clinically significant by the investigator
13. Body Mass Index (BMI) lower than 18 kg/m2 or greater than 35 kg/m2
14. In the opinion of the investigator, the subject is not suitable for the study
15. Any positive urine drug result or alcohol test at screening or admission, and/or a positive COVID-19 test performed at admission.
16. Any planned COVID-19 vaccination within a week of dosing through the duration of the trial
17. Currently a smoker or a nicotine user

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 hours
  Incidence and type of adverse events reported and observed
Cmax | 24 hours
  Maximum observed plasma concentrations
Tmax | 24 hours
  Time in hours to maximum concentration assessed over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Don Kellerman, PharmD, Study Director — Zosano Pharma Corporation
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No